CLINICAL TRIAL: NCT06584318
Title: Exploratory Study of the Impact of Intermittent Hypoxia Intervention on Patients With Colorectal Cancer
Brief Title: Exploratory Study of Intermittent Hypoxia Intervention on Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IH-CC
Record Dates: First submitted 2024-07-31; First posted 2024-09-04 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): Participants will receive 14 times intermittent hypoxia (oxygen concentration: 13%) intervention before the surgery.
  Interventions: Other: Intermittent hypoxia intervention

INTERVENTIONS:
Other: Intermittent hypoxia intervention — The intermittent hypoxia protocol refers to 6 cycles of 10 minutes hypoxia inhaling interval by 5 minutes normoxia, which is performed twice a day (at least 6 hours apart) in 7 days.

SUMMARY:
This study aims to explore the safety and efficacy of intermittent hypoxia intervention on patients with colorectal cancer.

DETAILED DESCRIPTION:
The hypoxic adaptive response is a form of acquired tolerance that occurs by activating internal cellular protective mechanisms and enhancing immune function.This technology was initially utilized in sports training and high-altitude medicine to enhance strength, endurance, and overall athletic performance, as well as to enhance the body's adaptation to high-altitude hypoxia. This technology was initially utilized in sports training and high-altitude medicine to enhance strength, endurance, and overall athletic performance, as well as to enhance the body's adaptation to high-altitude hypoxia.

Intermittent hypoxia (IH) refers to periodic hypoxic-normoxic training performed with brief exposure to hypoxia. Previous studies have found that short-term intermittent hypoxia can increase the sensitivity of hypoxia and reduce the severity of acute hypoxia injury, and alleviate acute hypoxia injury by reducing the inflammatory response caused by hypoxia. Intermittent hypoxia has been shown in our team's work to effectively inhibit colorectal cancer tumor progression in mice by enhancing immune cell function. This study aims to explore the safety and efficacy of IH in patients with colorectal cancer using a non-randomized self-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer between ages of 18 and 65 years.
* Colorectal cancer stage Ⅰ,Ⅱ.
* Subjects or their legally authorized representative can provide informed consent.

Exclusion Criteria:

* History of cardiovascular, cerebrovascular, dermatological, and hematological diseases.
* History of pulmonary, hepatic, kidney, dermatologic and hematologic diseases.
* History of pregnancy, hypertension, diabetes mellitus, obesity, sleep apnea and neurological disorders.
* History of substance abuse.
* Participating in other drug or medical device studies.
* History of organ transplantation, including allogeneic stem cell and immune cell transplantation.
* Recent severe infection within 4 weeks.
* Received cancer treatment, including chemotherapy and radiotherapy, within 4 weeks.
* Underwent major surgery within 28 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | During the 7-day treatment
  Adverse reactions included headache, vomiting, diarrhea, fatigue, dizziness and insomnia.

SECONDARY OUTCOMES:
Tumor Markers | The day before the 7-day treatment ; the day of surgery (1-7days post the treatment)
  Blood tumor markers will be detected by the immunochemiluminescence method.
Tumor Change | The day before the 7-day treatment ; the day of surgery (1-7days post the treatment)
  Tumor Change will be detected by tumor cell HIF-1α and HIF-2α through immunohistochemistry.
Cytokines | The day before the 7-day treatment ; the day of surgery (1-7days post the treatment)
  Cytokines will be detected by immune-related cytokines in peripheral blood.
Immune Cell Infiltration | The day before the 7-day treatment ; the day of surgery (1-7days post the treatment)
  Immune Cell Infiltration will be detected by observation of immune cell infiltration in tumor tissue.
Symptoms | The day before the 7-day treatment ; the day of surgery after the treatment;7 days after surgery
  It is evaluated by completing the follow-up form.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No